CLINICAL TRIAL: NCT04629417
Title: Measuring Adherence to Home Shoulder Physiotherapy With Artificial Intelligence
Acronym: SPARS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPARS2019
Record Dates: First submitted 2020-08-14; First posted 2020-11-16 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2024-07

CONDITIONS: Rotator Cuff Pathology
Keywords: Rehabilitation; Artificial Intelligence; Wearable Electronic Devices; Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Injured Worker Population (Experimental): Participants that have a confirmed rotator cuff pathology, and are undergoing physiotherapy at the Holland Centre for a work-related shoulder injury as part of the Working Condition Program.
  Interventions: Device: Smart Physiotherapy Activity Recognition System (SPARS)
- OHIP (funded) Patient Population (Active Comparator): Participants that have a confirmed rotator cuff pathology, and are undergoing physiotherapy at the Holland Centre as part of the Shoulder Program.
  Interventions: Device: Smart Physiotherapy Activity Recognition System (SPARS)

INTERVENTIONS:
Device: Smart Physiotherapy Activity Recognition System (SPARS) — Wearable smart watch that records inertial data such as (accelerometer, gyroscope magnetometer) while patients are performing physiotherapy exercises.

SUMMARY:
An important part of recovery for shoulder injuries, is sticking to the exercise regimen that is prescribed by a physiotherapist. Currently, there is no proper way to measure whether patients are correcting doing their prescribed exercises at home. Researchers at Sunnybrook have tested out a Smart Physiotherapy Recognition System (SPARS), which consists of a watch that patients can wear while they are performing their physiotherapy exercises. The watch aims to learn how the exercises are done correctly when worn during supervised physiotherapy sessions, and then to record and compare whether those same exercises are being done correctly in a home setting. The main objectives of this study aims to test whether the SPARS system can effectively measure whether physiotherapy exercises are being done properly when they are done without physiotherapist supervision. Secondly, to examine whether the recovery process after shoulder injuries is improved if patients perform the physiotherapy exercises correctly.

DETAILED DESCRIPTION:
A research assistant will conduct in-person data collection on 120 patients, by recording patients' exercises during their supervised physiotherapy sessions each week using the SPARS smart watch. Each patient will wear smart watch on their affected arm only when performing prescribed exercises, and the watch will start recording inertial sensor data once the patient puts the watch on. The injured worker population will be recruited from referrals made to the Sunnybrook Working Condition Program (WCP) at the Holland Centre for a work-related shoulder injury. The patient population that is being funded by OHIP, will be recruited from referrals Sunnybrook Shoulder and Upper Extremity Program. Data collection will be collected at baseline (at time of informed consent), and at each supervised physiotherapy session during the course of a patient's treatment. A research assistant will be required to attend a minimum of one supervised physiotherapy session for each patient every two weeks, and record exercise type and technique, alongside the inertial data collection, based on feedback from the treating physiotherapist. Follow-up outcomes such as surveys and shoulder testing will be done at 6 weeks, monthly at a maximum of 3 months (OHIP-patients) and 5 months (WSIB) patients, final treatment session (if different than maximum amount), and 1 year after.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females over the age of 18
2. Be diagnosed with rotator cuff tendinosis, shoulder impingement syndrome or a rotator cuff tear
3. Will be undergoing planned conservative management
4. Be able to participate in home physiotherapy exercises

Exclusion Criteria:

1. Upper extremity neurological deficit
2. Have had a previous failed surgery on the shoulder that is currently being treated
3. Undergoing simultaneous treatment for both shoulders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2024-02-16 (Actual)

PRIMARY OUTCOMES:
Physiotherapy participation (smart watch inertial data) | Up to 3-5 months
  Watch will begin recording inertial sensor data when it is put on during supervised and home physiotherapy exercises, and will stop recording when it is removed.

SECONDARY OUTCOMES:
Work status | Up to 1 year
  Clinical and return to work outcome data Full-time, part-time, off-work, modified or regular duties
Numeric Pain Rating Scale (NPRS) | Up to 1 year
  Scale range: 0 to 10 (whole number integers). Higher scores represent more pain.
The Disabilities of the Arm, Shoulder and Hand (DASH) Score | Up to 1 year
  Self administered questionnaire to self rate upper extremity disability and symptoms. Comprises of a 30-item disability/symptom scale, and higher scores represent more symptoms/disability.
Strength testing | Up to 12 weeks
  Rotator cuff strength testing using manual muscle testing as well as strength testing with a dynamometer
Shoulder active range of motion | Up to 12 weeks
  Measured by handheld goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Robin Richards, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Holland Orthopaedic & Arthritic Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Littlewood C, Bateman M, Clark D, Selfe J, Watkinson D, Walton M, Funk L. Rehabilitation following rotator cuff repair: a systematic review. Shoulder Elbow. 2015 Apr;7(2):115-24. doi: 10.1177/1758573214567702. Epub 2015 Jan 29. PMID 27582966
- [Background] Thomson S, Jukes C, Lewis J. Rehabilitation following surgical repair of the rotator cuff: a systematic review. Physiotherapy. 2016 Mar;102(1):20-8. doi: 10.1016/j.physio.2015.08.003. Epub 2015 Sep 8. PMID 26510584
- [Background] Jack K, McLean SM, Moffett JK, Gardiner E. Barriers to treatment adherence in physiotherapy outpatient clinics: a systematic review. Man Ther. 2010 Jun;15(3):220-8. doi: 10.1016/j.math.2009.12.004. Epub 2010 Feb 16. PMID 20163979
- [Background] Faber M, Andersen MH, Sevel C, Thorborg K, Bandholm T, Rathleff M. The majority are not performing home-exercises correctly two weeks after their initial instruction-an assessor-blinded study. PeerJ. 2015 Jul 21;3:e1102. doi: 10.7717/peerj.1102. eCollection 2015. PMID 26244112
- [Background] Bollen JC, Dean SG, Siegert RJ, Howe TE, Goodwin VA. A systematic review of measures of self-reported adherence to unsupervised home-based rehabilitation exercise programmes, and their psychometric properties. BMJ Open. 2014 Jun 27;4(6):e005044. doi: 10.1136/bmjopen-2014-005044. PMID 24972606
- [Background] Burns DM, Leung N, Hardisty M, Whyne CM, Henry P, McLachlin S. Shoulder physiotherapy exercise recognition: machine learning the inertial signals from a smartwatch. Physiol Meas. 2018 Jul 23;39(7):075007. doi: 10.1088/1361-6579/aacfd9. PMID 29952759
- [Background] Beaton DE, Katz JN, Fossel AH, Wright JG, Tarasuk V, Bombardier C. Measuring the whole or the parts? Validity, reliability, and responsiveness of the Disabilities of the Arm, Shoulder and Hand outcome measure in different regions of the upper extremity. J Hand Ther. 2001 Apr-Jun;14(2):128-46. PMID 11382253
- [Background] Staples MP, Forbes A, Green S, Buchbinder R. Shoulder-specific disability measures showed acceptable construct validity and responsiveness. J Clin Epidemiol. 2010 Feb;63(2):163-70. doi: 10.1016/j.jclinepi.2009.03.023. Epub 2009 Aug 14. PMID 19683414